CLINICAL TRIAL: NCT04425486
Title: Parents' Knowledge, Attitudes &Awareness Toward Pediatric Dentistry
Brief Title: Parents' Knowledge Toward Pediatric Dentistry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rana mohamed sabry ali mohamed el roby, doctor Rana, Cairo University
Other Study IDs: 200
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Parents' Knowledge

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the Parents' Knowledge, Attitudes &Awareness toward Pediatric Dentistry.

DETAILED DESCRIPTION:
Primary teeth are the valuable assets of a child. In children, milk teeth/primary teeth play a vital role for eating, phonetics and esthetics. Primary teeth are also essential in the development of the mouth. They maintain the arch length within the jaw and provide guides for the eruption pathway of the permanent teeth.

Problems in primary teeth in the form of pain and swelling can cause distress to the child, leading to inability to chew or speak properly and even may affect the appearance of a child. Premature loss of primary teeth can cause an earlier eruption of permanent successors and interfere with the harmony of adult dentition resulting in crowding caused by shifting and or drifting of the teeth toward the extraction space. Moreover, psychological, morphological and functional problems may result from premature loss of primary teeth.

Most parents are unaware of the role a pediatric dentist plays in their child's life, and the importance of dental visits at an early age is underestimated as most believe that the milk teeth are going to exfoliate and it not worth paying much attention to. Even if a parent is recommended to take the child to a pediatric dentist, many may not consider doing the same since awareness of importance of primary teeth is less.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 3 years- 12 years.
* Children with no previous dental treatment.
* Healthy children without any systemic diseases.

Exclusion Criteria:

* Refusal of participations.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parents of children(aged 3-12 years)
Sampling Method: Non-Probability Sample
Enrollment: 369 (Estimated)
Dates: Start 2020-10-05 (Estimated); Primary Completion 2021-07-05 (Estimated); Study Completion 2021-08-08 (Estimated)

PRIMARY OUTCOMES:
Parents' Knowledge, Attitudes &Awareness toward Pediatric Dentistry | after 3 months
  Data will be collected through a questionnaire for assessing parent's knowledge, attitudes &awareness toward pediatric dentistry.